CLINICAL TRIAL: NCT06958653
Title: Gamified Digital Balance Assessment for Older Adults in Community Settings: Development, Validation, and User Experience Evaluation in a Mixed Methods Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Jianan Zhao, Principle investigator, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Balance assessment tool
Record Dates: First submitted 2025-04-17; First posted 2025-05-06 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2024-01

CONDITIONS: ELDERLY PEOPLE; Fall Prevention; Digital Health

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Active Comparator): Participants in the control group used Brief-BESTest to assess their balance ability
  Interventions: Device: Brief-BESTest assessment
- Experimental group (Active Comparator): Participants in the experimental group uses the Gamified Digital Balance Assessment to assess their balance ability
  Interventions: Device: Digital balance assessment tool
- Gamified group (Experimental): The GDBA builds upon the digitalized Brief-BESTest by incorporating evidence-based gamification elements designed to enhance motivation and engagement among older adults. The gamification design was guided by self-determination theory, which posits that autonomy, competence, and relatedness are key drivers of intrinsic motivation, and by recent systematic reviews on gamification for older adult health interventions.
  Interventions: Device: Gamified Digital Balance Assessment (GDBA)

INTERVENTIONS:
Device: Brief-BESTest assessment — Uses the traditional Brief-BESTest to assess the balance ability of the participants.
  Arms: Control group
Device: Digital balance assessment tool — Uses the digital balance assessment tool, which is the digitalized Brief-BESTest, to assess their balance ability.
  Arms: Experimental group
Device: Gamified Digital Balance Assessment (GDBA) — The GDBA builds upon the digitalized Brief-BESTest by incorporating evidence-based gamification elements designed to enhance motivation and engagement among older adults. The gamification design was guided by self-determination theory, which posits that autonomy, competence, and relatedness are key drivers of intrinsic motivation, and by recent systematic reviews on gamification for older adult health interventions.
  Arms: Gamified group

SUMMARY:
The study was conducted in two sequential phases to evaluate the reliability and user experience of a GBDA tailored for community-dwelling older adults.

Phase 1: Reliability of digitalized Brief-BESTest assessment In the first phase, participants performed a single balance assessment session, during which both the clinician-administered Brief-BESTest and the digitalized Brief-BESTest were scored concurrently. This approach enabled direct comparison between clinical and automated assessments under identical task conditions.

Testing was conducted in a controlled indoor setting featuring a 1 m × 1 m, 10 cm-thick EVA foam mat (35D density) and safety handrails on three sides. Prior to the assessment, participants completed a baseline questionnaire collecting demographic data (age, sex), anthropometric measurements (height, weight), and fall history (past 12 months). Written informed consent was obtained from all participants.

During the assessment, a certified physical therapist delivered standardized verbal instructions and rated each task using the validated Brief-BESTest rubric (maximum score = 24). Simultaneously, the digitalized Brief-BESTest system recorded participants' movements using a monocular 4K camera and calculated scores via an algorithm that mirrors the original scoring criteria. The torso and joint movements were analyzed in real time, and balance scores were automatically computed.

To evaluate inter-rater reliability, a second trained clinician independently rated 20% of the sample. This concurrent scoring design ensured consistent task execution while enabling evaluation of inter-method reliability of the automated system's scoring against expert clinician judgment.

Phase 2: Impact of GBDA on User Experience The second phase involved a parallel group randomized controlled trial to assess the impact of gamification on user experience. Participants were randomly assigned (1:1) to either the control group (uses digitalized Brief-BESTest) or the experimental group (uses GDBA) through a simple coin-randomization method by a blinded researcher. Testing was conducted in a 1 m × 3 m evaluation zone equipped with front, side, and rear safety railings, and a centrally placed EVA foam pad (identical to Phase 1). The DBTS system included a display screen, a Logitech Brio 4K webcam (30 fps) for motion tracking, and a built-in speaker for voice prompts. A detachable, ergonomically designed user console-compliant with Chinese anthropometric standards-was mounted on the front railing for interface navigation (see Figure 2).

In the control group, participants performed balance tasks following pre-recorded verbal instructions from a certified physical therapist. In the experimental group, tasks were presented via the GDBA interface, which included animated avatars, voice guidance, progress indicators, and real-time performance feedback. Each participant completed one practice trial per task to minimize learning effects, followed by the formal assessment. A 2-minute seated rest period was provided between tasks to reduce fatigue.

Immediately following the assessment, participants completed self-report measures on perceived exertion, intrinsic motivation, and intention for continued use. They then participated in a brief semi-structured interview exploring their perceptions of system usability and engagement. All interviews were audio-recorded and transcribed for thematic analysis. Participants received a nominal compensation (USD $10 equivalent) upon study completion.

ELIGIBILITY:
Inclusion Criteria:

* aged 60 or older,
* living independently,
* able to walk with or without an assistive device (without external help),
* willing and able to provide informed consent.

Exclusion Criteria:

* conditions that impede walking (e.g., hip fractures, lower limb amputations, hemiparesis),
* medications causing dizziness or affecting balance (e.g., psychotropic drugs),
* self-reported cardiovascular, pulmonary, neurological, musculoskeletal, or mental disorders,
* severe fatigue or pain,
* severe uncorrected vision or hearing impairments that may affect their ability to interact with the digital system

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2025-04-20 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-09-20 (Actual)

PRIMARY OUTCOMES:
Perceived physical exertion | Through intervention completion, an average of 10 mins
  Perceived physical exertion was measured using the Borg Rating of Perceived Exertion (RPE) Scale, ranging from 6 ("no exertion") to 20 ("maximal exertion"). Participants verbally reported their RPE immediately after completing all balance tasks to reflect overall physical demand and fatigue during the assessment. This measure provided insight into the tolerability and physical burden of the assessment procedures.
Motivational engagement | Through intervention completion, an average of 10 mins
  Motivational engagement was evaluated using the Intrinsic Motivation Inventory (IMI), a validated tool employing a 7-point Likert scale (1 = "not at all true," 7 = "very true") . Three subscales were analyzed: Interest/Enjoyment (assesses task engagement and inherent enjoyment of the activity); Perceived Competence (measures self-perceived ability and confidence in performing the tasks); Pressure/Tension (evaluates task-related stress and anxiety). Subscale scores were calculated as the mean of item responses, with higher scores indicating greater enjoyment, competence, or pressure, respectively. The IMI has demonstrated good internal consistency and construct validity in older adult populations
Intention to continue use | Through intervention completion, an average of 10 mins
  Intention to continue use was assessed through both quantitative and qualitative methods. Quantitatively, participants rated their likelihood of using the system again on a single-item 7-point Likert scale (1 = "very unlikely," 7 = "very likely") immediately following the assessment. Qualitatively, semi-structured interviews explored factors influencing future use intentions. Interview questions included: "Would you consider using this system regularly for balance checking? Why or why not?" and "What features would encourage you to use this system more often?" Interviews lasted 3-5 minutes, were audio-recorded with permission, transcribed verbatim, and analyzed using Braun and Clarke's six-phase thematic analysis framework.

OTHER OUTCOMES:
Balance confidence | Prior to the intervention
  Balance confidence was assessed as baseline variable using the Activities-specific Balance Confidence (ABC) scale (0-100%); for reporting consistency, ABC scores were normalized to a 0-1 scale by dividing by 100 and were collected immediately after the assessment session. Higher scores indicate greater balance confidence.
Balance ability | Through intervention completion, an average of 10 mins
  Balance ability was assessed using the Brief-BESTest, a validated clinical tool comprising eight tasks across six domains of postural control: biomechanical constraints, stability limits/verticality, anticipatory postural adjustments, postural responses, sensory orientation, and stability in gait. Each task is scored on a 0-3 scale (0 = inaccurate performance, 3 = normal performance), yielding a total score of 0-24, with higher scores indicating better balance.

CONTACTS AND LOCATIONS:
Locations (1):
- Hongqi Community, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
Information might be shared after publication.